CLINICAL TRIAL: NCT02087995
Title: Effectiveness and Safety Study of the Dexcom G4 Platinum With Modified Algorithm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PTL901100
Record Dates: First submitted 2014-02-03; First posted 2014-03-14 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2015-08

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Continuous Glucose Monitoring System (Experimental): Single-Arm, CGM Device Glucose challenge performed during a clinic session to obtain accuracy data for the CGM system compared to a venous reference measurement
  Interventions: Device: Continuous Glucose Monitoring

INTERVENTIONS:
Device: Continuous Glucose Monitoring — A prescribed clinic session day for participating subjects.
  Other Names: CGM System; G4 Platinum CGM System; Dexcom G4 CGM System

SUMMARY:
To establish the performance of the Dexcom G4 Platinum with a Modified Algorithm continuous monitoring system when compared to a laboratory reference measurement.

DETAILED DESCRIPTION:
A study to evaluate the performance of a modification to the G4 Platinum CGM system in adults with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years or older
* Diagnosis of Type 1 diabetes or Type 2 diabetes on Intensive Insulin Therapy (ITT)
* Willing to participate in a clinic session

Exclusion Criteria:

* Use of Acetaminophen during study period
* Pregnancy
* Hematocrit (HCT) <35% (females) and 38% (males)
* Dialysis, history of cardiovascular disease, epilepsy, severe migraines in the past 6 months, adrenal disease, syncope, significant hypoglycemia unawareness, or a history of severe hypoglycemia within the last 6 months.
* Any condition that, in the opinion of the Investigator, would interfere with their participation in the study or pose and excessive risk to study staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andy Balo, Study Chair — DexCom, Inc.
Locations (3):
- United States (3):
  - John Muir Physician Network Clinical Research, Concord, California
  - AMCR Institute, Escondido, California
  - Diablo Clinical Research, Inc., Walnut Creek, California

REFERENCES:
- [Derived] Peyser TA, Nakamura K, Price D, Bohnett LC, Hirsch IB, Balo A. Hypoglycemic Accuracy and Improved Low Glucose Alerts of the Latest Dexcom G4 Platinum Continuous Glucose Monitoring System. Diabetes Technol Ther. 2015 Aug;17(8):548-54. doi: 10.1089/dia.2014.0415. Epub 2015 May 11. PMID 25961446

RESULTS

PARTICIPANT FLOW:
Groups:
- Real Time Continuous Glucose Monitoring System: Real Time Continuous Glucose Monitoring System Wear over a 7 day period
Period: Overall Study
Arm/Group | Real Time Continuous Glucose Monitoring System
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Type 1 and Type 2 diabetes patients
Arm/Group | Real Time Continuous Glucose Monitoring System
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years old] | 46.7 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 48
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Agreement of the Continuous Glucose Monitoring System Glucose Values Comparing to a Laboratory Reference, Yellow Sprint Instrument (YSI) Measurement.
Description: The percentage of CGM system values that are within 20% of the reference value for YSI glucose levels > 80 mg/dL or within 20 mg/dL at the reference glucose levels < 80 mg/dL.
Time Frame: 7-day wear period
Population: For the demographic and other baseline characteristic information, data from all 51 enrolled subjects was summarized.
Measure: Number; unit: Units analyzed% matched pairs w/i %20/20
Arm/Group | Real Time Continuous Glucose Monitoring System
Number analyzed (Participants) | 51
Units analyzed% matched pairs w/i %20/20 | 93

ADVERSE EVENTS:
Time Frame: 7 days of continuous glucose monitoring system use.
Description: AEs assessed for all participants enrolled into the study
Arm/Group | Real Time Continuous Glucose Monitoring System
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 1/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real Time Continuous Glucose Monitoring System (N=51)
Blister, skin (Skin and subcutaneous tissue disorders) | 1 (1) — Skin blister from study procedures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No